CLINICAL TRIAL: NCT04360317
Title: Phase I Study to Evaluate the Maximum Tolerated Dose of the Combination of SH003 and Docetaxel in Patients With Solid Cancer
Brief Title: Safety of the Combination of SH003 and Docetaxel in Patients With Solid Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Gyu Ko, Prof., Kyunghee University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISEE_2018_SH003
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Combination of SH003 and Docetaxel

INTERVENTIONS:
Drug: Combination of SH003 and Docetaxel — Combination of SH003 and Docetaxel

SUMMARY:
The study is designed as a single Group, Dose Elevating trial which evaluates safety to confirm the final maximum tolerated dose by the combination of oral administration of SH003 to docetaxel administered patients.

Firstly, 3 subjects is recruited and administered for 21 days for the starting dose of 2,400 mg / day. If no DLT occurs, raise the dose to a secondary dose of 3,600 mg / day. If DLT occurs, additional 3 subjects are recruited and administered for 2,400mg / day. After, If two or more of the six subjects shows DLT, stop the capacity increase, whereas if DLT occurs in less than 1 person, increase the dose to 3,600 mg / day. Next, 3 subjects is recruited and administered for 21 days for a dose of 3,600 mg / day. If no DLT occurs, raise the dose to 4,800 mg / day. If DLT occurs, 3 subjects are additionally recruited and administered for 3,600 mg / day. After, If two or more of the six subjects shows DLT, stop the capacity increase, whereas if DLT occurs in less than 1 person, increase the dose to 4,800 mg / day. Finally, 3 subjects is recruited and administered for a dose of 4,800 mg / day. If no DLT occurs, complete the study. If DLT occurs, additional 3 subjects are recruited and administered for 4,800mg / day and complete the study after observation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged above 19 years
2. Patients with histologically or cytologically confirmed lung cancer or breast cancer for which standard curative measures do not exist or are no longer effective
3. Patients who have not received chemotherapy, radiotherapy or surgery within the last 4 weeks and no residual toxicity associated with the previous treatment (Grade 1 or higher adverse event according to Common Terminology Criteria for Adverse Events (CTCAE) ver 5.0 from the National Cancer Institute (NCI)
4. ECOG Performance Status ≤ 2
5. Life expectancy estimated to be at least 12 weeks
6. Patients with the ability to swallow tablets
7. Patients with measurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
8. Patients with proper organ function as follows i. Bone marrow function: haemoglobin ≥8 g/dL, absolute neutrophil count ≥1,500/uL, and platelets ≥ 100,000/uL ii. Liver function: total bilirubin, aspartate aminotransferase (AST), or alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN) (if patients with liver metastasis, ≤ 5 times the ULN) iii. Renal function: Serum creatinine ≤ 1.5 times the ULN or creatinine clearance according to the Cockroft-Gault equation ≥ 60 ml/min
9. No possibility of pregnancy if the participant is female (over 60 years of age, without menstruation for more than one year, or underwent hysterectomy or bilateral oophorectomy). If there is a possibility of pregnancy, pregnancy test should be conducted prior to participation in the study to prove that it is not pregnancy
10. Patients who agree to use effective means of contraception during the trial and up to 8 weeks after final administration
11. Patients with the ability to understand the study and who are willing to sign a written informed consent document

Exclusion Criteria:

1. Patients undergoing any systemic therapy or regional therapy including radiotherapy, for the purpose of treating cancer
2. Participants with known hypersensitivity to any study drug component, including Astragalus membranaceus, Angelica gigas, Trichosanthes Kirilowii Maximowicz, and polysorbate 80
3. Patients with active infections requiring treatment (active hepatitis A, B, and C viruses, human immunodeficiency virus, tuberculosis)
4. Patients with history of human immunodeficiency virus infection
5. Patients with uncontrolled cardiovascular diseases (unstable angina, heart failure, myocardial infarction, hypertension that remains uncontrolled: 140/90 mm Hg or higher)
6. Patients with active cytomegalovirus infection within the past 4 weeks
7. Patients who have experienced major surgery on cerebrovascular disease such as acute coronary syndrome, stroke, etc., within the past year
8. pregnant or lactating females
9. Patient with metastatic encephalopathy with symptoms
10. Patients who have donated blood or participated in other clinical trials of medicine or medical devices within the past month
11. Patient underwent organ transplantation including allogenic stem cell transplantation
12. Patients with complications of infectious diseases
13. Patients with suspected fever caused by infection
14. Patients with substance abuse or any neurological, medical, psychological, or sociological conditions that could potentially interfere with their compliance to the study protocol or interpretation of study results
15. Patients who are judged inappropriate for the study by investigator
16. Patients who are judged to have lost their ability to consent due to accompanying disease such as dementia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | up to 4 weeks
  adverse event according to CTCAE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheon C, Ko SG. Phase I study to evaluate the maximum tolerated dose of the combination of SH003 and docetaxel in patients with solid cancer: A study protocol. Medicine (Baltimore). 2020 Sep 18;99(38):e22228. doi: 10.1097/MD.0000000000022228. PMID 32957363